CLINICAL TRIAL: NCT05117580
Title: Risk Reduction in Patients With Metabolic Syndrome Through Telemedicine-led Lifestyle Interventions
Brief Title: Telemedicine With Metabolic Syndrome
Acronym: METSZI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Szeged University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: TMED_METSZI_001
Record Dates: First submitted 2021-10-05; First posted 2021-11-11 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-10

CONDITIONS: Metabolic Syndrome; Life Style
Keywords: Telemedicine
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active group (Experimental): The active group get telemedicine devices, and lifestyle interventions.
  Interventions: Device: telemedicine lifestyle guidance
- Comparator Group (No Intervention): The comparator group get the evidence based treatment.

INTERVENTIONS:
Device: telemedicine lifestyle guidance — Telemedicine lifestyle advices are given during 3 months, based on telemonitoring system data.
  Arms: Active group

SUMMARY:
Investigation of the effect of a 3-month telemedicine-led lifestyle intervention on cardiovascular risk factors, functional indicators, in patients with metabolic syndrome.

DETAILED DESCRIPTION:
The patients are using mobile phone-based nutrition diary with heart rate monitoring watch (including activity meter) connected to a mobile phone with bluetooth technology worn on a wrist. These devices, and the weight scale, blood pressure monitor are connected with bluetooth to an IT system, that transmits and displays data from these devices. the patients are using the devices during 3 months, and get instructions about lifestyle.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 years and 75 years
* Presence of at least three of the following five risk factors (Metabolic Syndrome ATP III Criteria):

  1. waist width above 102 cm in men and 88 cm in women
  2. treated diabetes or blood sugar above 5.6 mmol / l
  3. treated hypertension or spontaneous blood pressure ≥ 130/85 mmHg
  4. fibrate treatment or triglyceride levels above 1.7 mmol / l
  5. blood HDL cholesterol levels below 1.03 mmol / l in men and 1.3 mmol / l in women

Exclusion Criteria:

* Low level of physical activity (less than 30 minutes a day)
* IT proficiency at least for basic use of mobile phones (answering / making voice calls).
* For women with childbearing potential, by definition, all women who are able to conceive physiologically use dual contraception
* Signing an informed consent.
* The subject communicates well with the investigator and is able to help understand and adhere to the requirements of the study plan.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Change of abdominal circumference | 3 months
  To investigate the effect of telemedicine-assisted lifestyle intervention on anthropometric parameters, with particular reference to the reduction of abdominal circumference in patients with metabolic syndrome.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4. | 3 months
  The safety of the device system
Impact of the system to the cardiovascular risk | 3 months
  In patients with metabolic syndrome, high cardiovascular risk, the impact of complex lifestyle interventions initiated in different environments and then telemedicine, including lifestyle and physical activity, on the known cardiovascular risk factors and functional indicators

CONTACTS AND LOCATIONS:
Locations (1):
- University of Szeged, Szeged, Hungary

IPD SHARING:
Plan to Share IPD: No